CLINICAL TRIAL: NCT02679846
Title: Safety of Antiepileptic Withdrawal in Long Term Video-EEG Monitoring
Acronym: SAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2014-852; 2014-A01460-47 (Other: ID-RCB)
Record Dates: First submitted 2016-02-08; First posted 2016-02-10 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Epilepsy
Keywords: withdrawal of antiepileptic drugs; monitoring VEEG; safety; adverse event; standardized protocol
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standardized protocol of AEDs withdrawal (Experimental): The standardized protocol of AEDs withdrawal will be implemented and applied to all inpatients
  Interventions: Other: Standardized protocol
- Current practice (No Intervention): Centers will continue their current practice

INTERVENTIONS:
Other: Standardized protocol — The standardized protocol of AEDs withdrawal will be implemented and applied to all inpatients
  Arms: Standardized protocol of AEDs withdrawal

SUMMARY:
SAVE is a stratified cluster-randomised controlled, parallel group, open-label trial, with Epileptic Monitoring Unit (EMU) as the units of randomisation and patients as the unit of analysis.

The focus of research is the management of AntiEpileptic Drugs (AEDs) withdrawal during long term Video EEG (VEEG) monitoring in patients with drug resistant seizures. This non-standardised medical practice, which aims at promoting the occurrence of seizures during the time limit of the monitoring period, exposes patients to significant risks which should be minimised by harmonisation of practice and a standardised protocol of AEDs withdrawal.

SAVE will assess the impact of a standardised protocol of AEDs withdrawal during long-term VEEG monitoring on the frequency of seizure-related serious adverse events occurring during these monitorings and on the ability to obtain VEEG recording of seizures within appropriate time limits.

10 of the 22 EMUs will be randomised to the group where the standardised protocol of AEDs withdrawal will be used systematically, while the other ten EMUs will continue their current non-standardised practice of AEDs withdrawal, and will serve as a control group.

The setting of the study will include a 6 months evaluation phase, prior to randomisation, during which the organisational characteristics, baseline EMUs' activity, current management of AEDs withdrawal, and rate of Serious Adverse Events (SAEs) of each participating center will be evaluated.

The standardised study protocol of AEDs withdrawal has been defined on the basis of a systematic review of all relevant publications in the field.

ELIGIBILITY:
Inclusion Criteria:

* Male or female suffering from drug-resistant epilepsy
* Age ≥ 6 years old
* Inpatient in one of the participating EMUs for recording seizure during long-term VEEG monitoring (≥ 48 hours)
* Patient who gave its written informed consent to participate to the study, or for children, whose minimum one of parents had given its written informed consent

Exclusion Criteria:

* Age < 6 years old
* Inpatient in one of the participating EMUs for performing short-term VEEG monitoring (<48 hours)
* Pregnant or breastfeeding woman

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1567 (Actual)
Dates: Start 2016-02-19 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who develop seizure-related serious adverse events during long-term VEEG monitoring | from date of inclusion until end of study (maximum 36 days)
  Proportion of patients who develop seizure-related serious adverse events during long-term VEEG monitoring, defined as the occurrence of one or more of the following events:
  * Convulsive or non-convulsive status epilepticus
  * 4-hour seizure cluster (≥ 3 seizures / 4 hours)
  * secondarily generalised seizure unusual for the patient (≤ 1/year)
  * vertebral compression
  * other fracture (including broken tooth)
  * post-ictal psychosis
  * post-ictal aspiration pneumonia
  * cardio-respiratory arrest
  * Any other seizure-related serious injury or adverse events

SECONDARY OUTCOMES:
Proportion of patients who develop each of the above seizure-related SAEs during long-term VEEG monitoring | from date of inclusion until end of study (maximum 36 days)
Proportion of patients who develop SAEs unrelated to the occurrence of a seizure, during long-term VEEG monitoring | from date of inclusion until end of study (maximum 36 days)
Proportion of patients who develop adverse events, including serious and non-serious adverse events, during long-term VEEG monitoring | from date of inclusion until end of study (maximum 36 days)
Delay between onset of monitoring and VEEG recording of the first seizure (in hours) | from date of inclusion until the first seizure (maximum 21 days)
Proportion of patients in whom at least one seizure will be recorded during the VEEG monitoring | from date of inclusion until the end of monitoring (maximum 21 days)
Proportion of patients in whom the duration of VEEG monitoring will extend beyond its initially scheduled time limits | from date of inclusion until the end of monitoring (maximum 21 days)
Duration of VEEG | from date of inclusion until the end of monitoring (maximum 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain RHEIMS, MD, Principal Investigator — Service de Neurologie Fonctionnelle et d'Epileptologie et Institut des Epilepsies
Locations (23):
- France (23):
  - Hôpital Nord, Amiens
  - CHU d'Angers, Angers
  - Hôpital R. Pellegrin, Bordeaux
  - Hôpital HFME, Bron
  - Hôpital P. Wertheimer, Bron
  - Hôpital Général, Dijon
  - Hôpital Michallon, Grenoble
  - Hôpital R. Salengro, Lille
  - Hôpital de La Timone, Marseille
  - Hôpital G. de Chauliac, Montpellier
  - Hôpital Central, Nancy
  - Hôpital Pasteur, Nice
  - La Pitié Salpétrière, Paris
  - Hôpital Necker, Paris
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris
  - Hôpital Robert Debré, Paris
  - Hôpital Pontchaillou, Rennes
  - Hôpital Ch. Nicolle, Rouen
  - Hôpital Nord, Saint-Etienne
  - Hôpital Hautepierre, Strasbourg
  - La Teppe, Tain-l'Hermitage
  - Hôpital Paul Riquet, Toulouse
  - CHU Bretonneau, Tours